CLINICAL TRIAL: NCT05565963
Title: Effectiveness of VR Exercise Intervention on Functional Fitness and Quality of Life Among Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: litingwang_2
Record Dates: First submitted 2022-09-23; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Health Promotion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group. (Experimental): 12-week intervention, with a 12-week follow-up. Device:1 computer virtual reality online software and 3 large projectors were used to project videos on the wall in a wrap-around state.
  Interventions: Other: Virtual reality exercise intervention
- Control group. (No Intervention): No intervention with a 12 week follow-up.

INTERVENTIONS:
Other: Virtual reality exercise intervention — The experimental group received VR exercise sessions for 75-90 minutes, twice a week for a duration of 12 weeks.
  Arms: Intervention group.

SUMMARY:
The aim of this study is to determine the effect of virtual reality-based exercise on the intervention and follow-up retention of functional fitness and quality of life among older adults.

DETAILED DESCRIPTION:
In a worldwide survey of fitness trends last 2021, Virtual Reality (VR) training recently took the top 10 spots. In fact, only a few studies were conducted on the retention of functional fitness and quality of life among older people. The main goal of this study was to assess the effects of virtual reality exercise on the functional fitness and quality of life of older adults after 12 weeks of intervention and another 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 65,
2. are able to perform daily activities,
3. with no past or current history of medical situations found in the Physical Activity Readiness Questionnaire (PAR-Q).

Exclusion Criteria:

1. being less than 65 years of age,
2. being unfit to participate in the study as revealed by the PAR-Q.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test to specify that "a period change" is being assessed. | The time points for assessment were week 1 (pre-test), 13 (post-test), and 24 (follow-up).
  Senior Fitness Tests were to evaluate the functional fitness of older adults. The test has six items: back scratch (cm), chair sit-and-reach (cm), arm curl, chair stand (times), 2-minute step (times), and 8-foot starting distance (sec). The functional fitness (e.g., back scratch, chair-and-reach, arm curl, chair stand, 2-minute step) of higher scores means better functional fitness.
  The functional fitness (e.g., 8-foot starting distance) of higher scores means poorer functional fitness.
  This study is a measure to assess change between two-time points.
  (1)Change in functional fitness of older adults from 1-week baseline (pre-test) to 12 weeks (i.e., exercise intervention phase). (2) Discontinuation of exercise intervention at 13 (post-test) to 24 weeks (follow-up) and ongoing follow-up of older people's function fitness maintenance outcomes.
Quality of Life Test to specify that "a period change" is being assessed. | Measured at week 1 (pre-test), 13 (post-test), and 24 (follow-up).
  The WHOQOL-OLD is used to measure the quality of life of older adults. This questionnaire is comprised of 24 items divided into six domains, with each domain having four items. These domains include sensory abilities, autonomy, response to the past present, and future activities, social participation, response to death and dying, and response to intimacy. Responses were rated on a Likert scale, with a 1-5-point scale for each item. The result with the highest total score indicates a greater quality of life.
  This study is a measure to assess changes between two-time points.
  (1) Change in self-perceived quality of life from 1-week baseline (pre-test) to 12 weeks (i.e., exercise intervention phase). (2) Discontinuation of exercise intervention at 13 (post-test) to 24 weeks (follow-up) and ongoing follow-up of older people's self-perceived quality of life maintenance outcomes.

SECONDARY OUTCOMES:
Body mass index (BMI) | Measured at week 1(pre-test).
  Measure older adults of height by attaching cloth ruler tape to the wall (units of measurement: cm). The weight of the elderly is measured using commercially available electronic weighing machines. (weight and height will be combined to report BMI in kg/m2).
International Physical Activity Questionnaire (IPAQ-LV). | Measured at week 1(pre-test).
  Physical activity was chosen through the Taiwanese version of the IPAQ-LV. Results were determined by first understanding how much total time was spent on physical activity. This was then multiplied by the frequency of the activity (i.e., per week and per day). The purpose of this was to evaluate the difference in physical activity of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Hsien Lee, Study Director — Research Ethics Committee, National Taiwan University, Taiwan
Locations (1):
- NTNU, Taipei, Taiwan